CLINICAL TRIAL: NCT01072006
Title: Top-Down Executive Control in TBI, PTSD and Combined TBI/PTSD
Brief Title: Top-Down Executive Control in Traumatic Brain Injury (TBI), PTSD and Combined
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Other Study IDs: D7031-W
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: PTSD; TBI (Traumatic Brain Injury)
Keywords: TBI (Traumatic Brain Injury); PTSD; fMRI; attention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control Group: Control group without traumatic brain injury (TBI) or post-traumatic stress disorder (PTSD)
- PTSD Group: PTSD (not TBI)
- TBI Group: TBI (no PTSD)
- TBI+PTSD Group: Combined TBI history and PTSD

SUMMARY:
This research investigates processes involved with one being able to focus on relevant information and ignore non-relevant information in veterans with PTSD and those with a history of traumatic brain injury. In addition, this study evaluates whether there is an additive effect of having both PTSD and history of TBI on ability to focus attention and inhibit distracting information.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) and PTSD both are characterized by deficits in attention, yet it is unclear as to whether this is related to an inability to focus on relevant information or ignore non-relevant information. History of TBI and PTSD are common to returning soldiers from OEF/OIF and thus is highly relevant to veteran health care. It is unclear how TBI and PTSD separately, and together, affect one's ability to focus attention versus inhibit distracting stimuli. This research investigates this issue by use of a working memory paradigm with functional magnetic resonance imaging (fMRI) that entails the subject being instructed to ignore some stimuli and remember other stimuli resulting in discrete biomarkers of (1) task-related enhancement of neural processes as well as (2) suppression of task-irrelevant neural processes. In this way, the specific aspect of attention in TBI and PTSD will be elucidated in addition to exploring whether PTSD and TBI have an additive, or even synergist, effect when combined.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be between 18 and 40 years of age.
* In order to be included in the mTBI group, participants must have sustained between 1 and 3 mild TBIs. The criteria for TBI will be consistent with what the VA currently uses (i.e., American Congress of Rehabilitative Medicine).
* More specifically, patients will have sustained a traumatically induced physiologic disruption of brain function as indicated by at least one of the following:

  * any period of loss of consciousness,
  * any loss of memory for events immediately before or after the accident,
  * any alteration in mental status at the time of the accident, and
  * focal neurologic deficits.
* Additional criteria for TBI include:

  * TBI must have been sustained during OEF or OIF and
  * TBI must consist of less than 30 minutes loss of consciousness, posttraumatic amnesia of less than 1 hour, and no positive CT/MRI findings.
* For PTSD group inclusion, psychiatric diagnoses will be established via the PTSD Clinical Checklist- Military (PCL-M) and the Clinician Administered PTSD Scale (CAPS).
* For PTSD/mTBI group inclusion, the above criteria must be met for both PTSD and mTBI.
* Control subjects will be OEF/OIF veterans with a history of exposure to combat without current or previous diagnosis of PTSD and no history of TBI.

Exclusion Criteria:

* Subjects who meet diagnostic criteria for drug abuse/dependence over the past year will be excluded.
* Individuals will be excluded if they have neurological confounds (e.g., baseline history of a CNS opportunistic infection, CNS neoplasm, neurosyphilis, current seizure disorder, demyelinating diseases), learning disorder, or current psychiatric disorders involving psychosis (schizophrenia, bipolar disorder with psychosis).
* Patients will also be excluded from the study if they are claustrophobic or are taking cardiovascular medications as these are contraindications for fMRI.
* All 4 subject groups will be matched for age and education.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: OEF/OIF Veterans enrolled in the Northern California Health Care System
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana V. Baldo, PhD, Principal Investigator — Martinez Outpatient Clinic and Community Living Center, Martinez, CA
Locations (1):
- Martinez Outpatient Clinic and Community Living Center, Martinez, CA, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sozda CN, Muir JJ, Springer US, Partovi D, Cole MA. Differential learning and memory performance in OEF/OIF veterans for verbal and visual material. Neuropsychology. 2014 May;28(3):347-352. doi: 10.1037/neu0000043. Epub 2013 Nov 18. PMID 24245926

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VANCHCS clinic recruitment 2011-2015
Pre-assignment Details: This was not a clinical trial so there was no random assignment to groups. Rather, patients fell into distinct groups based on their clinical history (e.g., history of TBI or PTSD or both or neither).
Period: Overall Study
Arm/Group | Control Group | PTSD Group | TBI Group | TBI+PTSD Group
Started | 14 | 5 | 0 | 11
Completed | 14 | 5 | 0 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | PTSD Group | TBI Group | TBI+PTSD Group | Total
Number analyzed (Participants) | 14 | 5 | 0 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 5 | 0 | 11 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (3.5) | 33.8 (7.2) |  | 28.8 (4.3) | 30.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 3
  Male | 12 | 5 | 0 | 10 | 27
Region of Enrollment [Number; unit: participants]
  United States | 14 | 5 |  | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Correlation
Description: Functional magnetic resonance imaging (fMRI) is used to measure neural activity in participants during attentional task, specifically measured as a bold signal change from rest to attention task. We then calculate the correlation between the bold signal (fMRI) and the PTSD CheckList questionnaire score. (The bold signal from fMRI indirectly reflects the brain's use of glucose, the brain's main energy source.) Correlations are reflected in an R-value, and R-values can range from 0-1, where 0 means there is no correlation (or relationship) between the two measures (here, the two measures are the fMRI brain signal and the PTSD score) and 1 means there is a perfect correlation between the two measures. A high correlation in this study would suggest that the more severe a patient's PTSD symptoms are, the harder their brain is having to work to accomplish the attention task. Separate correlations were analyzed for each group, and the overall R-value for each group is reported below.
Time Frame: These are chronic patients and controls who will only be tested at one time point, which corresponds to their entry into the study (after signing consent forms). Data collected at this single time point will be reported.
Measure: Number; unit: r-value
Arm/Group | Control Group | PTSD Group | TBI+PTSD Group
Number analyzed (Participants) | 14 | 5 | 11
r-value | .21 | .19 | .36

2. Secondary Outcome: Psychodiagnostic Testing: Post-traumatic Stress Disorder Check List (PCL) Measures the Level of Post-traumatic Stress Disorder (PTSD) Symptoms
Description: The PCL is a 17-item questionnaire that measures PTSD symptoms on a scale that ranges from 17-85 points. The total severity score is reported below. A higher score means a higher level of PTSD symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | PTSD Group | TBI Group | TBI+PTSD Group
Number analyzed (Participants) | 14 | 5 | 0 | 11
units on a scale | 27.2 (9.4) | 56.6 (11.2) |  | 60.4 (12.3)

3. Secondary Outcome: Neuropsychological Testing (Wechsler Test of Adult Reading)
Description: This test provides an estimate of pre-morbid IQ, which is important to report so that the patient sample can be compared to other similar studies for comparable IQ level and so that pre-morbid IQ can be considered as a potential variable. There are 50 items that are each given a score of 1, so the range of scores is 0-50. The raw score is then converted into an estimated IQ score based on age and education. The scores reported below reflect this estimated IQ score, where normal IQ scores range from 75 as low average to 125 as high average.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | PTSD Group | TBI Group | TBI+PTSD Group
Number analyzed (Participants) | 14 | 5 | 0 | 11
units on a scale | 103.3 (5.7) | 95.2 (7.9) |  | 102.1 (8.9)

ADVERSE EVENTS:
Arm/Group | Control Group | PTSD Group | TBI Group | TBI+PTSD Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/5 | 0/0 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/5 | 0/0 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No